CLINICAL TRIAL: NCT00862992
Title: Phase II Study of MP-214 in Patients With Schizophrenia (Exploratory Study)
Brief Title: Safety, Pharmacokinetics and Efficacy Study of MP-214 in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A002-A3
Record Dates: First submitted 2009-03-15; First posted 2009-03-17 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia; antipsychotics; dopamine D3/D2 antagonist
MeSH Terms: conditions — Schizophrenia | interventions — cariprazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Cariprazine 3 mg
- 2 (Experimental)
  Interventions: Drug: Cariprazine 6 mg
- 3 (Experimental)
  Interventions: Drug: Cariprazine 12.5 mg

INTERVENTIONS:
Drug: Cariprazine 3 mg
  Other Names: Cariprazine(INN); RGH-188
  Arms: 1
Drug: Cariprazine 6 mg
  Arms: 2
Drug: Cariprazine 12.5 mg
  Arms: 3

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics and efficacy of 3 fixed doses of MP-214 orally administered once daily to patients with schizophrenia. MP-214 tablets will be administered to patients starting at an initial dose, followed by up-titration to a fixed dose (low, medium or high) for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting DSM-IV-TR criteria for schizophrenia
* PANSS total score <= 120 during the observation period
* Patients who have been treated with oral antipsychotics within 4 weeks before informed consent
* Patients whose consent is obtained from themselves in written form

Exclusion Criteria:

* Patients who have defined as any mental disorder other than "Schizophrenia" based on the criteria of DSM-IV-TR
* History of drug or alcohol abuse
* Concurrent Parkinson's disease
* History of, or concurrent spastic disorders like epilepsy, cerebrovascular disease, anuresis or adynamic(= paralytic) ileus, malignant syndrome, diabetes, hepatic disorder
* Patients who exhibit abnormalities on Physical Examination, have abnormal vital signs, ECG, or clinical laboratory values
* Current cataract during the observation period
* History of shock or anaphylactoid symptoms to drugs

The information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teruhiko Higuchi, President, Study Chair — National Center of Neurology and Psychiatry
Locations (1):
- Hoyu Hospital, Kure, Hiroshima, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg
Started | 12 | 10 | 12
Completed | 9 | 9 | 9
Not Completed | 3 | 1 | 3
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg | Total
Number analyzed (Participants) | 12 | 10 | 12 | 34
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0
  >=18 and =<30 years | 2 | 2 | 2 | 6
  >=31 and =<40 years | 2 | 4 | 3 | 9
  >=41 and =<55 years | 6 | 3 | 5 | 14
  >55 years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 4 | 14
  Male | 6 | 6 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Event and Adverse Drug Reaction
Time Frame: Up to 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg
Number analyzed (Participants) | 12 | 10 | 12
Participants
  Number of Participants With Adverse event | 9 | 9 | 11
  Number of Participants With Adverse drug Reaction | 5 | 6 | 10

2. Secondary Outcome: Maximum Plasma Concentration of Unchanged MP-214, M7 (Desmethyl Cariprazine) and M6 (Didesmethyl Cariprazine) at Day 14
Time Frame: Pre-dose, 3, 4, 6, 8, 24, 48, 72, 96 and 168 hours post-dose of Day 14.
Population: Of the 34 participants, 7 subjects who prematurely discontinued during the titration period, 1 subject used prohibited concomitant medication and 1 subject did not take the test product on Day 12 of the fixed-dose period were excluded from the pharmacokinetic analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg
Number analyzed (Participants) | 9 | 8 | 8
ng/mL
  Unchanged MP-214 | 9.19 (3.47) | 19.43 (4.80) | 36.39 (8.53)
  M7 (desmethyl cariprazine) | 3.14 (1.26) | 5.83 (1.87) | 11.37 (3.00)
  M6 (didesmethyl cariprazine) | 13.79 (5.74) | 28.08 (14.52) | 54.99 (14.97)

3. Secondary Outcome: Time to Maximum Plasma Concentration of Unchanged MP-214, M7 (Desmethyl Cariprazine) and M6 (Didesmethyl Cariprazine) at Day 14
Time Frame: Pre-dose, 3, 4, 6, 8, 24, 48, 72, 96 and 168 hours post-dose of Day 14.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg
Number analyzed (Participants) | 9 | 8 | 8
hour
  Unchanged MP-214 | 3.71 (0.99) | 3.48 (1.11) | 3.22 (0.45)
  M7 (desmethyl cariprazine) | 5.25 (1.99) | 5.10 (1.94) | 4.36 (1.80)
  M6 (didesmethyl cariprazine) | 4.79 (2.23) | 5.37 (2.14) | 5.22 (2.08)

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last of Unchanged MP-214, M7 (Desmethyl Cariprazine) and M6 (Didesmethyl Cariprazine) at Day 14
Time Frame: Pre-dose, 3, 4, 6, 8, 24, 48, 72, 96 and 168 hours post-dose of Day 14.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg
Number analyzed (Participants) | 9 | 8 | 8
ng*hr/mL
  Unchanged MP-214 | 298.36 (128.04) | 522.38 (194.61) | 1017.96 (419.24)
  M7 (desmethyl cariprazine) | 135.25 (64.80) | 232.38 (113.31) | 437.64 (131.76)
  M6 (didesmethyl cariprazine) | 1884.24 (785.73) | 3397.12 (2395.44) | 5950.73 (1928.05)

5. Other Pre Specified Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 14 (Last Observation Carried Forward; LOCF)
Description: PANSS score is a 30-item rating scale to assess both the positive and negative symptom syndromes of patients with schizophrenia. Each item is scored on a 7-point scale, from 1 (absent) to 7 (extreme). The PANSS total score of the 30 PANSS items ranges from 30 to 210. High scores indicate greater severity of symptoms.
Time Frame: at baseline, and on Day 14 or a last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg
Number analyzed (Participants) | 12 | 10 | 12
units on a scale | -0.2 (12.8) | -0.6 (15.6) | -3.9 (10.8)

6. Other Pre Specified Outcome: Change From Baseline in the Clinical Global Impression-Severity (CGI-S) Score at Day 14 (Last Observation Carried Forward; LOCF)
Description: CGI-S is a 7-point scale to assess the global severity of the participant's illness. CGI-S scores range from 1 (normal, not ill at all) to 7 (extremely ill).
Time Frame: at baseline, and on Day 14 or a last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg
Number analyzed (Participants) | 12 | 10 | 12
units on a scale | 0.3 (0.8) | -0.1 (0.9) | -0.1 (0.7)

7. Other Pre Specified Outcome: The Clinical Global Impression-Improvement (CGI-I) Score at Day 14 (Last Observation Carried Forward; LOCF)
Description: CGI-I is a 7-point scale to assess the global improvement of the participant's illness relative to baseline. CGI-I scores range from 1 (very much improved) to 7 (very much worse).
Time Frame: on Day 14 or a last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg
Number analyzed (Participants) | 12 | 10 | 12
units on a scale | 4.1 (1.3) | 3.7 (1.2) | 3.8 (1.1)

ADVERSE EVENTS:
Arm/Group | Cariprazine 3 mg | Cariprazine 6 mg | Cariprazine 12.5 mg
Serious Adverse Events (participants affected / at risk) | 3/12 | 1/10 | 2/12
Other Adverse Events (participants affected / at risk) | 9/12 | 9/10 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine 3 mg (N=12) | Cariprazine 6 mg (N=10) | Cariprazine 12.5 mg (N=12)
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Neuroleptic malignant syndrome (Nervous system disorders) | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 2 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine 3 mg (N=12) | Cariprazine 6 mg (N=10) | Cariprazine 12.5 mg (N=12)
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 3
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 2 | 0
Feeling abnormal (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2
Thirst (General disorders) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 3 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Blood prolactin increased (Investigations) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1
Blood urine present (Investigations) | 1 | 0 | 0
Glucose urine present (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 3
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Akathisia (Nervous system disorders) | 1 | 1 | 3
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 1 | 1
Sleep paralysis (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 3 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Poor personal hygiene (Social circumstances) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other